CLINICAL TRIAL: NCT04158388
Title: Effects of Nutritional Strategies or Manual Therapies on Physical and Psychological Parameters in Women With Fybromyalgia.
Brief Title: Effects of Nutritional Strategies or Manual Therapies in Women With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Assistant Professor, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UA-2019-04-10
Record Dates: First submitted 2019-10-14; First posted 2019-11-08 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Fibromyalgia
Keywords: micronutrients; nutrition; therapy; chronic disease
MeSH Terms: conditions — Fibromyalgia; Chronic Disease | interventions — Tryptophan; Magnesium; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EXPERIMENTAL DIET GROUP (Experimental)
  Interventions: Other: Mediterranean-diet enriched with a higher dose of tryptophan and magnesium
- CONTROL GROUP (Other)
  Interventions: Other: Isocaloric diet
- EXPERIMENTAL MASSAGE GROUP (Experimental): That group received moderate pressure digital manual therapy.
  Interventions: Other: Manual therapy
- EXPERIMENTAL PLACEBO GROUP (Experimental): That group was treated with a US (in off mode) without conductive gel. Placebo group.
  Interventions: Other: Placebo therapy

INTERVENTIONS:
Other: Mediterranean-diet enriched with a higher dose of tryptophan and magnesium — That gruop eaten at both breakfast and dinner from walnuts (3-5 units), as food with high values of tryptophan and magnesium
  Arms: EXPERIMENTAL DIET GROUP
Other: Isocaloric diet — That group eaten isocaloric diet plan based on Mediterranean diet.
  Arms: CONTROL GROUP
Other: Manual therapy — That group received moderate pressure digital manual therapy.
  Arms: EXPERIMENTAL MASSAGE GROUP
Other: Placebo therapy — That group was treated with a US (in off mode) without conductive gel.
  Arms: EXPERIMENTAL PLACEBO GROUP

SUMMARY:
The study had two objectives. The first main aim was to analyze the effects of tryptophan and magnesium-enriched Mediterranean diet on psychological variables (trait anxiety, self-image, mood state, eating disorders) and sleep effects in women with fibromyalgia. Our hypothesis, based on previous positive effects of tryptophan and magnesium supplementation by separate in this population, may improve psychological health and regulate sleep disruptions. The second aim was to assess the effectiveness of a manual therapy technique performed with moderate digital pressure in fibromyalgia patients on the variables of fatigue, pain, sleep, anxiety and mood. It was done to provide an alternative treatment to pharmacological therapies for fibromyalgia patients and to provide new evidence on the effects of manual therapy in fibromyalgia patients.

ELIGIBILITY:
Inclusion Criteria:

- Women aged 40-60 with fibromialgia (officially diagnosed).

Exclusion Criteria:

* Women used analgesics, vitamins containing supplements, and or other drugs for the treatment of fibromyalgia symptoms, or participation in other clinical trials.
* Women that be performing simultaneously to this study some other physical therapy or physical exercise treatment. Not having sufficient cognitive level to collaborate in the study or not having the possibility of attending the established sessions.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | 4 - 16 weeks
  Sleep Quality assessment: Athenas Insomnia Scale.
Anxiety trait | 4 - 16 weeks
  Anxiety trait assessment: Stay Trait Anxiety Inventory.
Mood state | 4 - 16 weeks
  Mood state assessment: Profile of Mood State inventory.
Fatigue severity | 4 - 16 weeks
  Fatigue severity assessment: Fatigue Severity Scale
Pain perception | 4 - 16 weeks
  Pain perception assessment: Visual Analogical Scale
Sleep quality | 4 - 16 weeks
  Sleep quality assessment: Pittsburgh Sleep Quality Index

SECONDARY OUTCOMES:
Body composition | 4 - 16 weeks
  Body composition assessment trough bioimpedance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alicante, Alicante, San Vicente Del Raspeig, Spain